CLINICAL TRIAL: NCT00853957
Title: An 8-week Multicenter, Randomized, Double-blind, Active Control, Parallel Group Study to Evaluate the Efficacy and Safety of Aliskiren Administered in Combination With Amlodipine (150/5 mg, 300/10 mg) Versus Amlodipine Alone (5 mg, 10 mg) in African American Patients With Stage 2 Hypertension
Brief Title: Efficacy and Safety of Aliskiren Administered in Combination With Amlodipine Versus Amlodipine Alone in African American Patients With Stage 2 Hypertension
Acronym: AACESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100AUS01
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension
Keywords: Hypertension; African Americans; Aliskiren; Amlodipine; Systolic blood pressure; Diastolic blood pressure; Stage II; Combination
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren/Amlodipine (Experimental): Aliskiren/Amlodipine 150 mg/5 mg titrated to 300 mg/10 mg
  Interventions: Drug: Aliskiren/Amlodipine
- Amlodipine (Active Comparator): Amlodipine 5mg titrated to 10 mg
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren/Amlodipine — Aliskiren/Amlodipine 150 mg/5 mg titrated to 300 mg/10 mg
  Arms: Aliskiren/Amlodipine
Drug: Amlodipine — Amlodipine 5 mg titrated to 10mg
  Arms: Amlodipine

SUMMARY:
The purpose of the study is to evaluate the BP-lowering efficacy of the combination of aliskiren and amlodipine, as initial therapy, compared to amlodipine monotherapy in African American patients with Stage II hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of African American background; self identified
* Patients with stage 2 hypertension defined as MSSBP ≥ 160 mmHg and < 200 mmHg at Visit 5 (randomization

Exclusion Criteria:

* Office blood pressure measured by cuff (MSDBP ≥ 110 mmHg and/or MSSBP ≥ 200 mmHg)
* Patients on 4 or more antihypertensive medications.
* Patients with uncontrolled hypertension (MSSBP >180 mmHg) taking more than 1 antihypertensive medication at Visit 1
* Refractory hypertension, defined as, unresponsive to triple drug therapy at the maximum dose of each drug, one of which must be a diuretic, and not at blood pressure goal (140/90 mmHg). Therapy with a fixed dose combination of two active substances represent two drugs.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Evidence of a secondary form of hypertension, including but not limited to any of the following:

  * coarctation of the aorta
  * hyperaldosteronism
  * unilateral or bilateral renal artery stenosis
  * Cushing's disease
  * polycystic kidney disease
  * pheochromocytoma
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of angioedema due to usage of an ARB or ACE inhibitor.
* History of hypertensive encephalopathy, cerebrovascular accident, transient ischemic attack, heart failure (NYHA Class II-IV), coronary bypass graft surgery (CABG), percutaneous coronary intervention (PCI), unstable angina pectoris, or myocardial infarction in the last 12 months

Other protocol defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (9):
- United States (9):
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Oxon Hill, Maryland
  - Investigative Site, Detroit, Michigan
  - Investigative Site, Trenton, New Jersey
  - Investigative Site, Brooklyn, New York
  - Investigative Site, Springfield Gardens, New York
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Milwaukeee, Wisconsin

REFERENCES:
- [Derived] Weinberger MH, Izzo JL Jr, Purkayastha D, Weitzman R, Black HR. Comparative efficacy and safety of combination aliskiren/amlodipine and amlodipine monotherapy in African Americans with stage 2 hypertension and obesity or metabolic syndrome. J Am Soc Hypertens. 2011 Nov-Dec;5(6):489-97. doi: 10.1016/j.jash.2011.08.005. Epub 2011 Sep 17. PMID 21925996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Started | 220 | 223
Completed | 206 | 204
Not Completed | 14 | 19
Not completed — Adverse Event | 9 | 3
Not completed — Unsatisfactory therapeutic effect | 0 | 2
Not completed — Subject withdrew consent | 4 | 5
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol deviation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Amlodipine | Amlodipine | Total
Number analyzed (Participants) | 220 | 223 | 443
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (9.33) | 52.4 (10.57) | 52.8 (9.97)
Age, Customized [Number; unit: participants]
  <55 years | 123 | 127 | 250
  ≥55 years | 97 | 96 | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 115 | 238
  Male | 97 | 108 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: To compare the change from baseline in mean sitting systolic blood pressure (msSBP) after 8 weeks of treatment with a combination of aliskiren and amlodipine treatment regimen (150/5 mg, 300/10 mg) versus an amlodipine treatment regimen (5 mg, 10 mg) in African American patients with Stage 2 hypertension.
Time Frame: Baseline, 8 weeks
Population: Full analysis set, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 220 | 222
mm Hg | -33.1 (14.53) | -27.8 (13.45)

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: To compare the change from baseline in mean sitting diastolic blood pressure (msDBP) after 8 weeks of treatment with a combination of aliskiren and amlodipine treatment regimen (150/5 mg, 300/10 mg) versus an amlodipine treatment regimen (5 mg, 10 mg).
Time Frame: Baseline, 8 weeks
Population: Full analysis set, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 220 | 222
mm Hg | -13.7 (9.60) | -10.4 (9.08)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure (BP) Control (<140/90 mmHg)
Description: Cumulative percentage of patients achieving BP control (<140/90 mmHg)for both treatment arms was calculated. Cumulative refers to achieving blood pressure control before or at the corresponding visit. If achieving blood pressure control occurred more than once, only the first occurrence was counted.
Time Frame: 8 weeks
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 206 | 204
Percentage of participants | 71.4 | 57.4

4. Secondary Outcome: Percentage of Responders (Patients With MSSBP < 140 mmHg or Decrease From Baseline of Greater Than or Equal to 20 mmHg)
Description: Cumulative percentage of responders (Responders are defined as patients with MSSBP <140 mmHg or a decrease from baseline ≥20 mmHg) during 8 weeks of treatment was calculated. Cumulative refers to achieving blood pressure control before or at the corresponding visit. If achieving blood pressure control occurred more than once, only the first occurrence was counted.
Time Frame: 8 weeks
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 206 | 204
Percentage of participants | 92.3 | 86.5

5. Secondary Outcome: Change From Baseline in MSSBP at Week 1 and 4
Description: Compare the change from baseline in MSSBP at week 1 and 4
Time Frame: Baseline, 1 and 4 weeks
Population: Full analysis set, Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 215 | 219
mm Hg
  Baseline to Week 1 | -20.5 (12.53) | -18.2 (13.01)
  baseline to Week 4 | -30.9 (13.30) | -27.3 (13.58)

6. Secondary Outcome: Percentage of Patients With Peripheral Edema by Visit
Description: Cumulative percentage of patients with peripheral edema was calculated. 'Cumulative' refers to patients with peripheral edema before or at the corresponding visit. If peripheral edema occurred more than once, only the first occurrence was counted. Peripheral edema is the swelling of tissues due to the accumulation of fluids. Peripheral edema was assessed by investigators during physical examination.
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Number analyzed (Participants) | 220 | 223
Percentage of participants
  Week 1 | 1.4 | 1.3
  Week 4 | 4.1 | 5.8
  Week 8 | 6.8 | 8.5

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Aliskiren/Amlodipine | Amlodipine
Serious Adverse Events (participants affected / at risk) | 1/220 | 1/223
Other Adverse Events (participants affected / at risk) | 25/220 | 31/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Amlodipine (N=220) | Amlodipine (N=223)
Angina unstable (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Amlodipine (N=220) | Amlodipine (N=223)
Oedema peripheral (General disorders) | 17 | 20
Headache (Nervous system disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.